CLINICAL TRIAL: NCT00910117
Title: Phase II Study of Nimotuzumab Plus PF as Induction Chemotherapy in Patients With Locally Advanced HNSCC
Brief Title: Induction Chemotherapy With Nimotuzumab in Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNTG 09-01
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Head and Neck Cancer
Keywords: HNSCC; induction chemotherapy; nimotuzumab
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — nimotuzumab; CF regimen; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nimotuzumab (Experimental): nimotuzumab plus PF regimen
  Interventions: Drug: nimotuzumab; Drug: PF regimen (cisplatin and 5-FU)

INTERVENTIONS:
Drug: nimotuzumab — nimotuzumab 400 mg d1
  Other Names: h-R3
Drug: PF regimen (cisplatin and 5-FU) — cisplatin 75 mg/m2 d1 and 5-FU 750 mg/m2/d CIV d1-5
  Other Names: PF

SUMMARY:
The aim of the study is to evaluate the role of nimotuzumab in the neo-adjuvant setting in patients with locally advanced HNSCC. The hypothesis is that the response would be increased with the combination of nimotuzumab and cisplatin and fluorouracil (PF) regimen.

DETAILED DESCRIPTION:
Induction chemotherapy followed by radiotherapy is the standard treatment for patients with unresectable HNSCC. However, the role of induction chemotherapy remains uncertain for resectable disease. Therefore, we plan to perform a phase II study to evaluate it, focusing on radiographic and pathologic response after induction chemotherapy. Moreover, a new EGFR monoclonal antibody (nimotuzumab) is incorporated with PF regimen. The hypothesis is the addition of nimotuzumab would improve the response without remarkably increase the toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-70 years old
* ECOG performance status 0-1
* Histologically confirmed and potentially resectable locally advanced (T2-4, N0-3, M0) HNSCC
* Adequate organ function

Exclusion Criteria:

* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection
* Previous serious cardiac disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
overall response rate | 6 weeks

SECONDARY OUTCOMES:
pathologic complete response | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China